CLINICAL TRIAL: NCT03593525
Title: A Randomized Controlled Trial of Symptom Screening by Children With Cancer and Feedback to Providers
Brief Title: SPARK Symptom Screening and Feedback to Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Pediatric Oncologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB: 000061139
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Oncology; Quality of Life
Keywords: Pediatric Oncology; Randomized Control Trial; Symptom Screening; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPARK Intervention (Experimental): Participants will complete symptom screening using SPARK once daily on a study-supplied iPad. For inpatients, daily reminders to complete SSPedi will appear on the iPad. Reports will be available to the child at any time. For outpatients, clinical research associates will provide the iPad in person daily and reports may be viewed at those encounters. The intervention is daily symptom screening with provision of reports to the healthcare team. Severe symptoms will result in email alerts. More specifically, SSPedi reports will be printed daily and provided in the patient chart. On days 1 and 3, an alert will be emailed to the physician providing direct medical care if any symptom is "a lot" or "extremely" bothersome (score 3 or 4 on 0-4 scale). Reports and alerts will have links to SPARK-housed CPGs.
  Interventions: Other: SPARK
- Standard of Care Arm (No Intervention): Participants randomized to the control arm will not complete daily symptom screening. They will complete SSPedi on days 1 and 5 to obtain the primary outcome. Health care providers will not be notified of their SSPedi scores and no symptom reports or symptom alerts will be generated.

INTERVENTIONS:
Other: SPARK — see above
  Arms: SPARK Intervention

SUMMARY:
Supportive care Prioritization, Assessment and Recommendations for Kids (SPARK) is a web-based application which builds upon the Symptom Screening in Pediatrics Tool (SSPedi) and consists of two components: (1) a symptom screening component centered on SSPedi; and (2) a supportive care clinical practice guideline (CPG) component. This proposal is a randomized controlled trial that compares daily completion of SSPedi via SPARK for 5 days with symptom feedback to healthcare providers compared with standard of care

DETAILED DESCRIPTION:
Participants will be children with cancer or hematopoietic stem cell transplantation (HSCT) recipients who are 8-18 years of age and who can understand English, and who are expected to be in hospital or in clinic daily for 5 days. This will be a multi-center RCT in which we will randomize children to either undergo daily symptom screening for 5 days with symptom reports provided to the healthcare team or standard of care. The primary outcome will be the self-reported day 5 total SSPedi score (range 0-60; higher worse). Secondary outcomes will be the day 5 self-reported individual symptom, pain and QoL scores, and documentation of symptoms and provision of interventions for symptoms over the 5 day trial. We will enroll 345 participants over 4 years from 7 Canadian centers

ELIGIBILITY:
Inclusion Criteria:

* 8 to 18 years of age
* Diagnosis of cancer or have received or about to receive HSCT
* Understand English
* Expected to be in hospital or clinic for 5 day

Exclusion Criteria:

* illness severity
* cognitive disability
* visual impairment

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 345 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Lillian Sung, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dupuis LL, Johnston DL, Dix D, McKillop S, Cook S, Crellin-Parsons N, Kulkarni K, Patel S, Vanan ML, Gibson P, Soman D, Kuczynski S, Tomlinson GA, Sung L. Symptom Screening for Hospitalized Pediatric Patients With Cancer: A Randomized Clinical Trial. JAMA Pediatr. 2025 Jan 1;179(1):11-18. doi: 10.1001/jamapediatrics.2024.4727. PMID 39535812

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled but excluded from assignment to study groups.
Period: Overall Study
Arm/Group | SPARK Intervention | Standard of Care Arm
Started | 176 | 169
Completed | 168 | 164
Not Completed | 8 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPARK Intervention | Standard of Care Arm | Total
Number analyzed (Participants) | 176 | 169 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 176 | 169 | 345
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 13.9 [8.0 to 18.4] | 13.6 [8.0 to 18.8] | 13.8 [8.0 to 18.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 74 | 150
  Male | 100 | 95 | 195
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Aboriginal | 1 | 3 | 4
  Arab or West Asian | 10 | 13 | 23
  Asian | 53 | 27 | 80
  Black or African American | 5 | 7 | 12
  Latin American | 4 | 5 | 9
  White | 78 | 92 | 170
  Other race or mixed race | 20 | 20 | 40
  Unknown or missing | 2 | 2 | 4
  Prefer not to say | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 176 | 169 | 345

OUTCOME MEASURES:

1. Primary Outcome: SSPedi (Symptom Screening in Pediatrics) Total Scores
Description: The primary outcome will be the self-reported total SSPedi score on day 5. The total SSPedi score is a validated measure that reflects the total burden of bothersome symptoms experienced. The total score is the sum of each of the 15 items' Likert scores which range from 0 (not at all bothered) to 4 (extremely bothered) to yield a total score that ranges from 0 (no bothersome symptoms) to 60 (worst bothersome symptoms).
Time Frame: Measure will be completed by all participants at baseline (day 1) and day 5±1 day.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPARK Intervention | Standard of Care Arm
Number analyzed (Participants) | 168 | 164
score on a scale
  SSPedi Baseline Total Scores | 13.2 (8.0) | 13.1 (8.2)
  SSPedi Day 5 Total Scores | 10.2 (7.4) | 12.7 (8.3)

2. Secondary Outcome: Number of Participants With a Self-reported Severely Bothersome SSPedi (Symptom Screening in Pediatrics) Score Per Symptom
Description: The subscale SSPedi score is a validated measure that reflects the burden of a bothersome symptom experienced. Each of the 15 symptoms assessed by the SSPedi questionnaire will serve as secondary outcomes. The subscale uses a Likert score that ranges from 0 (not at all bothered) to 4 (extremely bothered). The reported values represent the number of participants who had symptoms rated as severely bothersome, defined as a score of 3 or 4 on the subscale. Higher reported scores indicate a higher number of participants that reported the level of bother for that symptom as a 3 or a 4.
Time Frame: Measure will be completed by all participants on baseline (day 1) and day 5±1 day.
Measure: Count of Participants; unit: Participants
Arm/Group | SPARK Intervention | Standard of Care Arm
Number analyzed (Participants) | 168 | 164
Participants
  SSPedi: Feeling sad or dissapointed baseline | 18 | 11
  SSPedi: Feeling scared or worried baseline | 18 | 17
  SSPedi: Feeling cranky or angry baseline | 10 | 11
  SSPedi: Problems thinking or remembering things baseline | 11 | 8
  SSPedi: Changes in how your body or face look baseline | 16 | 15
  SSPedi: Feeling tired baseline | 55 | 54
  SSPedi: Mouth sores baseline | 12 | 9
  SSPedi: Headache baseline | 10 | 11
  SSPedi: Hurt or pain (other than headache) baseline | 24 | 24
  SSPedi: Tingly or numb hands or feet baseline | 10 | 5
  SSPedi: Throwing up or feeling like you may throw up baseline | 17 | 19
  SSPedi: Feeling more or less hungry than you usually do baseline | 40 | 30
  SSPedi: Changes in taste baseline | 24 | 19
  SSPedi: Constipation baseline | 16 | 10
  SSPedi: Diarrhea baseline | 15 | 11
  SSPedi: Feeling dissapointed or sad day 5 | 8 | 10
  SSPedi: Feeling scared or worried day 5 | 4 | 6
  SSPedi: Feeling cranky or angry day 5 | 8 | 16
  SSPedi: Problems with thinking or remembering things day 5 | 2 | 9
  SSPedi: Changes in how your body or face look day 5 | 9 | 18
  SSPedi: Feeling tired day 5 | 31 | 53
  SSPedi: Mouth sores day 5 | 9 | 12
  SSPedi: Headache day 5 | 8 | 8
  SSPedi: Hurt or pain day 5 | 15 | 22
  SSPedi: Tingly or numb hands or feet day 5 | 4 | 4
  SSPedi: Throwing up or feeling like you may throw up day 5 | 17 | 23
  SSPedi: Feeling more or less hungry than you usually do day 5 | 21 | 35
  SSPedi: Changes in taste day 5 | 14 | 18
  SSPedi: Constipation day 5 | 6 | 14
  SSPedi: Diarrhea day 5 | 8 | 11

3. Secondary Outcome: Faces Pain Scale-Revised
Description: Self-reported pain will be assessed using the Faces Pain Scale-Revised which consists of a series of horizontal faces that depict a neutral facial expression of no pain on the left and worst pain on the right. It has 6 faces and may be scored on a 0 to 10 scale in which higher numbers denote more pain.
Time Frame: Measure will be completed by all participants on day 1 (baseline) and day 5±1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPARK Intervention | Standard of Care Arm
Number analyzed (Participants) | 168 | 164
score on a scale
  Face Pain Scale-Revised score baseline | 1.6 (1.9) | 1.4 (1.9)
  Face Pain Scale-Revised score day 5 | 1.7 (2.1) | 1.4 (1.9)

4. Secondary Outcome: PedsQL (Pediatric Quality of Life) 3.0 Acute Cancer Module
Description: Self-reported QoL will be measured using the PedsQL 3.0 Acute Cancer Module. This measure is a multidimensional instrument that is reliable and valid in children with cancer. It assesses pain and hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance and communication. The self-report 7-day recall version will be used. The problems are rated from 0; never a problem to 4 if it is almost always a problem. They produce 8 domain scores ranging from 0 to 100, with higher scores denote better health.
Time Frame: Measure will be completed by all participants on day 1 (baseline) and day 5±1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPARK Intervention | Standard of Care Arm
Number analyzed (Participants) | 168 | 164
score on a scale
  PedsQL 3.0 Pain and hurt baseline | 66.5 (26.5) | 68.3 (26.5)
  PedsQL 3.0 Nausea baseline | 69.2 (22.2) | 71.6 (20.7)
  PedsQL 3.0 Procedural Anxiety baseline | 65.5 (29.4) | 63.8 (32.7)
  PedsQL 3.0 Treatment Anxiety baseline | 77.0 (25.7) | 78.6 (25.8)
  PedsQL 3.0 Worry baseline | 62.4 (26.9) | 62.9 (27.0)
  PedsQL 3.0 Cognitive problems baseline | 69.7 (21.3) | 70.1 (21.3)
  PedsQL 3.0 Perceived physical appearance baseline | 75.3 (24.4) | 75.4 (26.2)
  PedsQL 3.0 Communication baseline | 72.9 (22.7) | 75.1 (23.1)
  PedsQL 3.0 Pain and hurt day 5 | 73.1 (22.6) | 72.8 (26.1)
  PedsQL 3.0 Nausea day 5 | 69.2 (21.8) | 69.5 (31.8)
  PedsQL 3.0 Procedural anxiety day 5 | 69.5 (29.9) | 66.5 (31.8)
  PedsQL 3.0 Treatment anxiety day 5 | 80.5 (23.7) | 81.9 (23.5)
  PedsQL 3.0 Worry day 5 | 68.7 (26.2) | 69.1 (25.4)
  PedsQL 3.0 Cognitive problems day 5 | 74.2 (21.4) | 74.4 (21.3)
  PedsQL 3.0 Percieved physical appearance day 5 | 79.2 (22.6) | 78.2 (25.5)
  PedsQL 3.0 Communication day 5 | 76.4 (22.3) | 78.1 (21.2)

ADVERSE EVENTS:
Time Frame: Adverse event data collected while participants were on study (period of 5 days ± 1 day)
Arm/Group | SPARK Intervention | Standard of Care Arm
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/169
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/169
Other Adverse Events (participants affected / at risk) | 0/176 | 0/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT03593525/Prot_SAP_001.pdf